CLINICAL TRIAL: NCT05848544
Title: Efficacy of a Very Low Calories Ketogenic Diet in Obese Patients With Fibromyalgia or Symptomatic Knee Osteoarthritis
Acronym: KD-FM-OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KD-FM-OA
Record Dates: First submitted 2023-04-13; First posted 2023-05-08 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Fibromyalgia; Knee Osteoarthritis
MeSH Terms: conditions — Fibromyalgia; Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symptomatic knee osteoarthritis (Other): obese patients with symptomatic knee osteoarthritis eligible to a very low calories ketogenic diet
  Interventions: Dietary Supplement: Very low-calorie ketogenic diet for patients with symptomatic knee osteoarthritis
- obese patients with fibromyalgia (Other): obese patients with with fibromyalgia eligible to a very low calories ketogenic diet
  Interventions: Dietary Supplement: Very low-calorie ketogenic diet for patients with fibromyalgia

INTERVENTIONS:
Dietary Supplement: Very low-calorie ketogenic diet for patients with symptomatic knee osteoarthritis — A personalized very low-calorie ketogenic diet will be prepared for each patient by specialized dietitians using a combination of commercially-available ketogenic preparations and patient's handmade prepared meals
  Arms: Symptomatic knee osteoarthritis
Dietary Supplement: Very low-calorie ketogenic diet for patients with fibromyalgia — A personalized very low-calorie ketogenic diet will be prepared for each patient by specialized dietitians using a combination of commercially-available ketogenic preparations and patient's handmade prepared meals
  Arms: obese patients with fibromyalgia

SUMMARY:
Adult patients with fibromyalgia or symptomatic knee osteoarthritis and comorbid obesity eligible to a very low calories ketogenic diet will be enrolled in the pilot study

DETAILED DESCRIPTION:
the study will be conducted following different periods:

1. Free diet (for 4 weeks). After recruitment, the patient will enter "free diet phase" in which he/she will be asked to follow a normal free diet for 4 weeks. During this period, a nutritional interview will be carried out by a trained dietician who will elaborate a personalized diet and order the ketogenic products on the basis of patient's preferences.
2. very low calories ketogenic diet (for 8 weeks). After the free diet period, the patient will start the very low calories ketogenic regimen. At the beginning of this period a box with the commercial products necessary to cover the whole study period will be hand-delivered by a dietician that will instruct the patient on the correct use and storage.
3. Maintenance (for 12 weeks). After very low calories ketogenic diet phase, the patient will start maintenance period as described

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 65 years
* Body mass index ≥ 30 kg/m2
* Failed to achieve weight loss with standard low-calories diet
* Any of the following conditions:

BMI ≥ 35 kg/m2 Past diagnosis of type 2 diabetes without β-cell failure Hypertriglyceridemia (fasting triglycerides ≥ 150 mg/dL) or taking lipid-lowering medications Hypercholesterolemia (total cholesterol > 200 mg/dL) or taking lipid-lowering medications Past diagnosis of arterial hypertension or taking blood pressure-lowering medications Past diagnosis of non-alcoholic fatty liver disease Past diagnosis of heart failure class NYHA I-II Past history of myocardial infarction (> 12 months), stroke/minor stroke (> 12 months) Past diagnosis of carotid atherosclerosis Past diagnosis of polycystic ovary syndrome (PCOS) Past diagnosis of neurodegenerative disorders

* Fibromyalgia classified according to 2016 Revisions to the 2010/2011 European League Against Rheumatism/ American College of Rheumatology OR
* Symptomatic knee osteoarthritis

Exclusion Criteria:

* Age < 18 or > 65 years
* Currently pregnant or breastfeeding
* Past diagnosis of type 1 diabetes mellitus, latent autoimmune diabetes in adults, β-cell failure in type 2 diabetes mellitus, use of sodium/glucose cotransporter 2 inhibitors (risk for euglycemic diabetic ketoacidosis)
* Past diagnosis of kidney failure and moderate-to-severe chronic kidney disease, liver failure, hearth failure NYHA III-IV, respiratory failure
* Past diagnosis of unstable angina
* Recent stroke or myocardial infarction (< 12 months)
* Cardiac arrhythmias
* Past diagnosis of eating disorders and other severe mental illnesses, alcohol and substance abuse
* Active/severe infections
* 48 h prior to elective surgery or invasive procedures and perioperative period
* Past diagnosis of rare disorders: porphyria, carnitine deficiency, carnitine palmitoyltransferase deficiency, carnitine-acylcarnitine translocase deficiency, mitochondrial fatty acid β-oxidation disorders, pyruvate carboxylase deficiency
* Allergy to protein-preparations ingredients
* Past or current history of gallstones

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
efficacy of the very low-calorie ketogenic diet in patient with fibromyalgia | baseline, 8 weeks and 20 weeks
  change in Fibromyalgia Impact Questionnaire total score for fibromyalgia
efficacy of the very low-calorie ketogenic diet in patient with osteoarthritis | baseline, 8 weeks and 20 weeks
  change in Western Ontario total score for osteoarthritis

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Derived] Ciaffi J, Mancarella L, Pederzani G, Lisi L, Brusi V, Pignatti F, Ricci S, Vitali G, Faldini C, Ursini F. Efficacy, Safety, and Tolerability of a Very Low-Calorie Ketogenic Diet in Women with Obesity and Symptomatic Knee Osteoarthritis: A Pilot Interventional Study. Nutrients. 2024 Sep 24;16(19):3236. doi: 10.3390/nu16193236. PMID 39408203
- [Derived] Ciaffi J, Lisi L, Mari A, Mancarella L, Brusi V, Pignatti F, Ricci S, Vitali G, Stefanelli N, Assirelli E, Neri S, Naldi S, Faldini C, Ursini F. Efficacy, safety and tolerability of very low-calorie ketogenic diet in obese women with fibromyalgia: a pilot interventional study. Front Nutr. 2023 Jul 12;10:1219321. doi: 10.3389/fnut.2023.1219321. eCollection 2023. PMID 37502721

DOCUMENTS (1):
  • Study Protocol (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT05848544/Prot_000.pdf